CLINICAL TRIAL: NCT04785768
Title: Intravenous (IV) Patient Controlled Analgesia (PCA) With or Without Continuous Dose vs Oral Opioid to Maintain Analgesia for Severe Cancer Pain After Successful Hydromorphone Titration: a Multi-center, Phase Ⅲ ，Randomized Trial
Brief Title: IV PCA With or Without Continuous Dose vs Oral Opioid to Maintain Analgesia for Severe Cancer Pain After Successful Titration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYLT021/HMORCT09-3
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cancer Pain
Keywords: Orally; IV PCA with continuous + bolus dose; IV PCA with bolus-only dose
MeSH Terms: conditions — Cancer Pain | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCA with continuous + bolus dose (Experimental): （1）Intravenous PCA with hydromorphone after successful titration of 24 hours;（2）PCA hydromorphone with continuous infusion where dose/h was the total equianalgesic over the previous 24h divided by 24 and bolus dosage for breakthrough pain was 10%-20% of the total equianalgesic over the previous 24h；lockout time = 10 minutes；（3）Evaluate every 24 hours and PCA parameters were adjusted according to the dose of the previous day; (4)The treatment regimen was continued for 7 days.
  Interventions: Drug: Hydromorphone Hydrochloride Injection
- PCA with bolus-only dose (Experimental): （1）Intravenous PCA with hydromorphone after successful titration of 24 hours; (2)PCA hydromorphone with bolus-only where dosage was 10%-20% of the total equianalgesic over the previous 24h administrated as needed;（3）Evaluate every 24 hours and PCA parameters were adjusted according to the dose of the previous day; (4)The treatment regimen was continued for 7 days.
  Interventions: Drug: Hydromorphone Hydrochloride Injection
- Oral opioid (Active Comparator): （1）Swift to sustained-release morphine orally as background dose with immediate release morphine orally for breakthrough pain after successful titration of 24 hours；(2)Oral sustained-released morphine where total equianalgesic over the previous 24h/2×75% every 12h/day and immediate-release morphine for breakthrough pain was 10%-20% of the total equianalgesic over the previous 24h； (3)Evaluate every 24 hours and the dose for the next day is adjusted according to the dose of the previous day；(4)The treatment regimen was continued for 7 days.
  Interventions: Drug: Morphine Sulfate Sustained-release Tablets

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride Injection — Intravenous PCA with hydromorphone after successful titration of 24 hours.the PCA setting: 1) continuous dose (dose/hours) = the total dosage of hydromorphone in the previous 24 hours/24; 2) bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours; 3) lockout time = 10 minutes; 4）Evaluate every 24 hours and PCA parameters were adjusted according to the dose of the previous day.
  Arms: PCA with continuous + bolus dose
Drug: Hydromorphone Hydrochloride Injection — Intravenous PCA with hydromorphone after successful titration of 24 hours.the PCA setting: 1) continuous dose = 0; 2) bolus dose = 10-20% of the total dosage of hydromorphone in the previous 24 hours: 3) lockout time = 10 minutes; 4)Evaluate every 24 hours and PCA parameters were adjusted according to the dose of the previous day.
  Arms: PCA with bolus-only dose
Drug: Morphine Sulfate Sustained-release Tablets — Swift to sustained-release morphine orally as background dose with immediate release morphine orally for breakthrough pain after successful titration of 24 hours.
  Administration of morphine orally 1) Sustained-release morphine orally (dose/12 hours) = the total equianalgesic of the previous 24 hours/2×75% for day 1; 2）the total equianalgesic of the previous 24 hours/2 for day 2 ; 3）Evaluate every 24 hours and the dose for the next day is adjusted according to the dose of the previous day；4) Immediate release morphine orally = 10-20% of the total equianalgesic of the previous 24 hours;
  Arms: Oral opioid

SUMMARY:
Based on the previous HMORCT09-2, the results show that IV PCA for analgesia maintenance improvements control of severe cancer pain after successful titration. Therefore, a study is planned to further explore the difference of efficacy and safety between PCA with continuous + bolus dose versus bolus-only.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 to 80 years;
2. Histologically or cytologically confirmed malignant solid tumor;
3. Persistent severe cancer-related pain (≥7 at rest on the 11-point numeric rating scale [NRS], where 0=no pain and 10=excruciating pain) in the 24 hours before screening;
4. No radiotherapy to the painful area prior to randomization;
5. No radiotherapy, chemotherapy, hormone therapy, targeted therapy, or bisphosphonate therapy within 7 days before randomization;
6. Successful IPCA-HM titration within the past 24 hours;
7. No history of psychiatric disorders;
8. Ability to complete questionnaires;
9. Ability to correctly understand and follow medication guidance from doctors and nurses;
10. ECOG performance status ≤ 3;
11. Provided written informed consent. Exclusion Criteria

1) Patients with non-cancer-related pain; 2) Patients with paralytic ileus; 3) Patients with brain metastases; 4) Patients with hypersensitivity to morphine or hydromorphone; 5) Abnormal laboratory results: creatinine ≥ 2-fold of upper limit of normal (ULN) value, Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 2.5-fold of the ULN value (≥ 5-fold for subjects with liver metastasis or primary liver cancer), or Child-Pugh class C liver function; 6) Patients unable to take oral medication; 7) Patients with uncontrolled nausea or vomiting; 8) Prior use of hydromorphone, morphine, or PCA devices within 14 days before screening; 9) Use of monoamine oxidase inhibitor drugs (MAOID) within the two weeks before randomization; 10) Women who are pregnant, lactating, or planning to be pregnant within one month after the trial completion; 11) Patients who abuse alcohol; 12) Patients with any other medical condition or reason, in the investigator's judgment, that would make them unsuitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
3DNRS (3-day average Numeric Rating Scale) | up to 4 days
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain. NRS of 24 hours is assessed every day. 3DNRS is a sum of average NRS of Day 1 (D 1) to Day 3 divided by 3 (the day of titration is defined as D0, the first day after titration is defined as D1, the second day after titration is defined as D2, and so on).

SECONDARY OUTCOMES:
Daily avNRS score of days 1 to 6 | up to 7 days
  Daily average NRS pain score of days 1 to 6
Adverse events | up to 8 days
  assessed by NCI-CTCAE v5.0
Improvement in physical symptoms and overall well-being | up to 7 days
  assessed by Chinese version of the Edmonton Symptom Assessment System.
Patient Satisfaction Score | up to 7 days
  The satisfaction score of the patients to analgesia was evaluated by 10-point scale: 0 points for dissatisfaction, 10 points for very satisfied, the higher the score, the higher the satisfaction.
Daily equivalent morphine consumption | up to 7 days
  Daily equivalent morphine consumption
Number of patients with an average NRS pain score > 6 | up to 7 days
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain.
Number of patients with an average NRS pain score >3 | up to 7 days
  The Numerical Rating Scale (NRS, a score of 0 means no pain and 10 means the most severe) is used to assess the severity of pain.
Patient Satisfaction Score | up to 7 days
  from 0 to 10, with 0 = extremely unsatisfied and 10 = extremely satisfied
Maximum NRS (Days 1 to 6) | up to 7 days
  Maximum NRS score (Days 1 to 6)
Daily frequency and duration of breakthrough cancer pain | up to 7 days
  Daily frequency and duration of breakthrough cancer pain (defined as transient pain exacerbation [NRS ≥4])

CONTACTS AND LOCATIONS:
Overall Officials: Rong bo Lin, MD, Principal Investigator — Fujian Cancer Hospital,Department of Gastrointestinal Medical Oncology
Locations (1):
- China, Fujian, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized individual participant data and supporting clinical trial documents, including the study protocol, informed consent forms, and statistical analysis plan, will be available upon reasonable request to the corresponding author